CLINICAL TRIAL: NCT04732169
Title: Cannabidiol for Treatment Resistant Depression
Acronym: CBD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator decided not to do study, due to insufficient funding.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Matthew Macaluso, Bee McWane Reid Professor, Department of Psychiatry & Behavioral Neurobiology, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 300006618
Record Dates: First submitted 2021-01-13; First posted 2021-02-01 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: We plan to administer Epidiolex (CBD) or placebo in double blind, randomized, cross-over fashion.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epidiolex (cannabidiol) (CBD) (Active Comparator): During the first week after randomization, participants will receive 125mg of Epidiolex (CBD) or matching placebo taken twice daily (250mg/day). During the second week after randomization, the dosage will be increased to 250mg of Epidiolex or placebo taken twice daily (500mg/day) for one week. During the third week after randomization, the dosage will be increased to 500mg of Epidiolex (CBD) or matching placebo taken twice daily (1000mg/day). Participants will remain on 1000mg/day of Epidiolex (CBD) or matching placebo for four more weeks, at which point they will be stepped down to 500mg/day of Epidiolex (CBD) or placebo for one week, followed by 250mg/day of Epidiolex (CBD) or placebo for one week.
  Interventions: Drug: Active study drug ( oral CBD)
- Placebo (Placebo Comparator): During the first week after randomization, participants will receive 125mg of Epidiolex (CBD) or matching placebo taken twice daily (250mg/day). During the second week after randomization, the dosage will be increased to 250mg of Epidiolex or placebo taken twice daily (500mg/day) for one week. During the third week after randomization, the dosage will be increased to 500mg of Epidiolex (CBD) or matching placebo taken twice daily (1000mg/day). Participants will remain on 1000mg/day of Epidiolex (CBD) or matching placebo for four more weeks, at which point they will be stepped down to 500mg/day of Epidiolex (CBD) or placebo for one week, followed by 250mg/day of Epidiolex (CBD) or placebo for one week.
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: Active study drug ( oral CBD) — CBD in single dose syringes
  Arms: Epidiolex (cannabidiol) (CBD)
Drug: matching placebo — Placebo made with sesame oil flavored with strawberry flavoring in single dose syringes
  Arms: Placebo

SUMMARY:
With this study, the investigators will address the following scientific aims:

1. Demonstrate the antidepressant effects of CBD in human adults with treatment refractory MDD as measured by standard rating scales.
2. Confirm CBD's safety profile in human adult patients with MDD.

DETAILED DESCRIPTION:
Participants will be medically stable and historically failed to respond to one or more adequate trials of commercially available antidepressant drugs during the current depressive episodes. We plan to administer Epidiolex (CBD) or placebo in double blind, randomized, cross-over fashion to 10 depressed adults with MDD over 16 weeks. The study will use a cross-over design so that each participant serves as their own control. The dosage of CBD or placebo CBD will automatically be titrated up and down during the dosing period. Participants first randomized to CBD will automatically be tapered from CBD and switched to placebo CBD after eight weeks. Participants first randomized to placebo CBD will automatically have an equivalent reduction in placebo CBD and be switched to CBD after eight weeks. During the first week after randomization, participants will receive 125mg of CBD or placebo CBD taken twice daily (250mg/day). During the second week after randomization, the dosage will be increased to 250mg of CBD or placebo CBD taken twice daily (500mg/day) for one week. During the third week after randomization, the dosage will be increased to 500mg of CBD or placebo CBD taken twice daily (1000mg/day). Participants will remain on 1000mg/day of CBD or placebo CBD for four more weeks, at which point they will be stepped down to 500mg/day of CBD or placebo CBD for one week, followed by 250mg/day of CBD or placebo CBD for one week.

Study drug and matching placebo will be prepared by the UAB Investigational Pharmacy. Sesame oil will be used to create the placebo. Both the placebo and the active CBD will be flavored with strawberry flavoring. Study medications will be dispensed at weekly visits and each participant will be given 14 single dose syringes to be taken orally twice a day.

At screening participants will undergo a MINI interview, physical examination, and ECG, vital signs, HDRS-17, MADRS, CSSR-S, ATRQ, SF-36 and CGI-S. Laboratory assessment including CBC with differential, TSH with reflex T4, CMP, UA, and UDS will be done at screening.. At screening, the investigators will also administer the following self-report questionnaires to characterize reward sensitivity and other personality features relevant to anhedonia: Social Anhedonia Scale, the Motivation and Energy Inventory and the Physical Anhedonia Scale. The screening period will last up to one week, at which point subjects will present for a baseline randomization visit.

Participants will be seen on site weekly during the study. Drug effect will be measured using standard rating scales including the HDRS-17, MADRS, SF36, CSSR-S, CGI-I, CGI-S, which will be completed at each visit. The following scales will be completed at every other visit following the screening visit: Social Anhedonia Scale, the Motivation and Energy Inventory and the Physical Anhedonia Scale. At each study visit safety assessments including vital sign assessment and adverse event assessment will be completed. Subjects will also undergo physical examination and an ECG for safety during screening, after 8 weeks of treatment and at the end of 16 weeks of treatment. Laboratory assessment including CBD with differential, CMP, and UA will be done at the 8 week and 16 week visit.

To assess potential changes in cognition while on the study drug/placebo, three computerized tests of cognition will the administered at baseline, Week 8, and Week 16. The Relational & Item Specific Encoding task (RISE) will probe any potential neural abnormalities. The Probabilistic Learning Task will be used to examine neural circuits related to reward processing in major depression disorder. For the working memory task, participants will be shown two images with objects and asked to decide whether the two images differ or not.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old
2. Sufficient fluency in English to understand testing procedures and provide written informed consent
3. A Hamilton Depression Rating Scale total score greater than 18
4. A DSM 5 diagnosis of MDD based on the MINI.
5. No evidence of alcohol or other substance use disorder in the past 3 months
6. For females: no current pregnancy or lactation (women of reproductive potential must have a negative urine pregnancy test at screening).
7. Depressed patients who have failed at least one adequate antidepressant trial during the current depressive episode based on the ATRQ.

   Exclusion Criteria:
8. No diagnosis of other primary psychiatric disorder (defined in this case as being the main focus of treatment) as determined by the MINI, such as: bipolar disorder, personality disorders, psychotic disorders, post-traumatic stress disorder, obsessive-compulsive disorder, dissociative disorders, eating disorder, or cognitive task due to neurological conditions
9. Systolic blood pressure < 150 and/or diastolic blood pressure < 90 at screening
10. A QTc F< 480 as determined by an ECG
11. No post-partum state (being within 2 months of delivery or miscarriage)
12. Imminent suicide or homicide risk as determined by the investigator
13. No history of using prescription Epidiolex for any indication.
14. Not being treated with one of the following medications: benzodiazepines or other CNS depressants.
15. Not using concomitant medications that are moderate or strong CYP3A4 or CYP2C19 inhibitors.
16. None of the following clinically-significant medication condition or therapy that would preclude treatment with ketamine, to include: Recent myocardial infarction, unstable angina, malignant neoplasm in the past 6 months, immunosuppressive or corticosteroid therapy within the last month, with the following exceptions: any inhaled, intranasal, topical or vaginal corticosteroids are allowed, chemotherapy.
17. No clinically significant neurological disease based on medical history (e.g., epilepsy) or significant head injury.
18. Any of the following disorders: Rheumatoid arthritis; Lupus erythematosus; Autoimmune hepatitis; Autoimmune peripheral neuropathy; Autoimmune pancreatitis; Behcet's disease; Crohn's disease; Autoimmune glomerulonephritis; Grave's disease; Guillain-Barre syndrome; Hashimoto's thyroiditis; Autoimmune polymyositis or polymyalgia; Myasthenia gravis; Narcolepsy; Polyarteritis nodosa; Scleroderma; Sjogren's syndrome; Transverse myelitis; Wegener's granulomatosis; History of seizures (only childhood febrile seizures are allowed)
19. The presence of clinically significant laboratory findings in the opinion of the investigator including, but not limited to, clinically significant anemia or transaminase elevation.
20. If the UDS is positive, the subject would be excluded if, in the opinion of the investigator, the positive UDS meant the subject has an active substance use disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale- 17 | Baseline
  A semi-structured interview focusing on 17 symptoms of depression, range of scores 0-52 with 0 indicating no depression
Hamilton Depression Rating Scale- 17 | Week 8
  A semi-structured interview focusing on 17 symptoms of depressionrange of scores 0-52 with 0 indicating no depression,
Hamilton Depression Rating Scale- 17 | Week 16
  A semi-structured interview focusing on 17 symptoms of depression, range of scores 0-52 with 0 indicating no depression.

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale | Baseline
  A 10 item semi-structured interview focusing on symptoms of depression, range of scores 0-60, with 0 indicating no depression
Montgomery Asberg Depression Rating Scale | Week 8
  A 10 item semi-structured interview focusing on symptoms of depression, range of scores 0-60, with 0 indicating no depression
Montgomery Asberg Depression Rating Scale | Week 16
  A 10 item semi-structured interview focusing on symptoms of depression, range of scores 0-60, with 0 indicating no depression

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Macaluso, D.O., Principal Investigator — University ot Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share protocol, consent, SAP,and CRS. Do not plan to share IPD,
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 years
Access Criteria: Will share with public

REFERENCES:
- [Background] Greenberg PE, Fournier AA, Sisitsky T, Pike CT, Kessler RC. The economic burden of adults with major depressive disorder in the United States (2005 and 2010). J Clin Psychiatry. 2015 Feb;76(2):155-62. doi: 10.4088/JCP.14m09298. PMID 25742202
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Stewart JW, Nierenberg AA, Thase ME, Ritz L, Biggs MM, Warden D, Luther JF, Shores-Wilson K, Niederehe G, Fava M; STAR*D Study Team. Bupropion-SR, sertraline, or venlafaxine-XR after failure of SSRIs for depression. N Engl J Med. 2006 Mar 23;354(12):1231-42. doi: 10.1056/NEJMoa052963. PMID 16554525
- [Background] Linge R, Jimenez-Sanchez L, Campa L, Pilar-Cuellar F, Vidal R, Pazos A, Adell A, Diaz A. Cannabidiol induces rapid-acting antidepressant-like effects and enhances cortical 5-HT/glutamate neurotransmission: role of 5-HT1A receptors. Neuropharmacology. 2016 Apr;103:16-26. doi: 10.1016/j.neuropharm.2015.12.017. Epub 2015 Dec 19. PMID 26711860
- [Background] Silote GP, Sartim A, Sales A, Eskelund A, Guimaraes FS, Wegener G, Joca S. Emerging evidence for the antidepressant effect of cannabidiol and the underlying molecular mechanisms. J Chem Neuroanat. 2019 Jul;98:104-116. doi: 10.1016/j.jchemneu.2019.04.006. Epub 2019 Apr 27. PMID 31039391
- [Background] Gall Z, Farkas S, Albert A, Ferencz E, Vancea S, Urkon M, Kolcsar M. Effects of Chronic Cannabidiol Treatment in the Rat Chronic Unpredictable Mild Stress Model of Depression. Biomolecules. 2020 May 22;10(5):801. doi: 10.3390/biom10050801. PMID 32455953
- [Background] Shbiro L, Hen-Shoval D, Hazut N, Rapps K, Dar S, Zalsman G, Mechoulam R, Weller A, Shoval G. Effects of cannabidiol in males and females in two different rat models of depression. Physiol Behav. 2019 Mar 15;201:59-63. doi: 10.1016/j.physbeh.2018.12.019. Epub 2018 Dec 17. PMID 30571957
- [Background] Sales AJ, Fogaca MV, Sartim AG, Pereira VS, Wegener G, Guimaraes FS, Joca SRL. Cannabidiol Induces Rapid and Sustained Antidepressant-Like Effects Through Increased BDNF Signaling and Synaptogenesis in the Prefrontal Cortex. Mol Neurobiol. 2019 Feb;56(2):1070-1081. doi: 10.1007/s12035-018-1143-4. Epub 2018 Jun 4. PMID 29869197
- [Background] Cuttler C, Spradlin A, McLaughlin RJ. A naturalistic examination of the perceived effects of cannabis on negative affect. J Affect Disord. 2018 Aug 1;235:198-205. doi: 10.1016/j.jad.2018.04.054. Epub 2018 Apr 6. PMID 29656267
- [Background] McGuire P, Robson P, Cubala WJ, Vasile D, Morrison PD, Barron R, Taylor A, Wright S. Cannabidiol (CBD) as an Adjunctive Therapy in Schizophrenia: A Multicenter Randomized Controlled Trial. Am J Psychiatry. 2018 Mar 1;175(3):225-231. doi: 10.1176/appi.ajp.2017.17030325. Epub 2017 Dec 15. PMID 29241357